CLINICAL TRIAL: NCT03507686
Title: An Open-Label Safety Study of Retinal Gene Therapy for Choroideremia With Bilateral, Sequential Administration of Adeno-Associated Viral Vector (AAV2) Encoding Rab Escort Protein 1 (REP1)
Brief Title: A Safety Study of Retinal Gene Therapy for Choroideremia With Administration of BIIB111
Acronym: GEMINI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 273CH203; 2017-002395-75 (EudraCT Number)
Record Dates: First submitted 2018-03-07; First posted 2018-04-25 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-08

CONDITIONS: Choroideremia
Keywords: NightstaRx; NSR-REP1; CHM; Gene Therapy; AAV; REP1; Timrepigene Emparvovec
MeSH Terms: conditions — Choroideremia | interventions — Genetic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BIIB111 (Experimental): Participants will receive a single dose of sub-retinal injection of BIIB111 in each eye at Day 0 separated by an interval of <6 months, 6-12 months, or >12 months.
  Interventions: Drug: BIIB111

INTERVENTIONS:
Drug: BIIB111 — Administered as specified in the treatment arm.
  Other Names: Gene Therapy; AAV2-REP1

SUMMARY:
The objective of the study is to evaluate the safety of bilateral, sequential sub-retinal administration of a single dose of BIIB111 in adult male participants with Choroideremia (CHM).

DETAILED DESCRIPTION:
This study was previously posted by NightstaRx Ltd. In October 2020, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

1. Are willing and able to give informed consent for participation in the study to have both eyes treated.
2. Have documentation of a genetically-confirmed diagnosis of CHM.
3. Have active disease clinically visible within the macular region of both eyes.
4. Have a BCVA of ≥34 ETDRS letters (20/200 or better Snellen acuity) in both eyes, or in the untreated eye, if the other eye was previously treated with BIIB111*

   *If previously treated with BIIB111 in an antecedent study, participants may be eligible for participation following Sponsor approval.
5. For participants who received treatment with BIIB111 in an antecedent study, have biological samples available to complete an adequate immunology profile.

Key Exclusion Criteria:

1. Have a history of amblyopia or inflammatory disorder in either eye.
2. Are unwilling to use barrier contraception methods or abstain from sexual intercourse for a period of 3 months following treatment with BIIB111 in either eye.
3. Have had previous intraocular surgery performed within 3 months of the Screening Visit in either eye.
4. Have any other significant ocular or non-ocular disease/disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the results of the study or the participant's ability to participate in the study. This includes but is not limited to a potential participants:

   * with a contraindication to oral corticosteroid (e.g., prednisolone/prednisone)
   * with clinically significant cataract in either eye
   * who, in the clinical opinion of the Investigator, is not an appropriate candidate for sub-retinal surgery.
5. Have participated in another research study involving an investigational product in the past 12 weeks or received a gene/cell-based therapy at any time previously, except if treated within an antecedent study with BIIB111.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (6):
- United States (4):
  - Research Site, Miami, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
- Research Site, Paris, France
- Research Site, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] MacLaren RE, Audo I, Fischer MD, Huckfeldt RM, Lam BL, Pennesi ME, Sisk R, Gow JA, Li J, Zhu K, Tsang SF. An Open-Label Phase II Study Assessing the Safety of Bilateral, Sequential Administration of Retinal Gene Therapy in Participants with Choroideremia: The GEMINI Study. Hum Gene Ther. 2024 Aug;35(15-16):564-575. doi: 10.1089/hum.2024.017. Epub 2024 Jul 27. PMID 38970425
- [Derived] Davis JL. The Blunt End: Surgical Challenges of Gene Therapy for Inherited Retinal Diseases. Am J Ophthalmol. 2018 Dec;196:xxv-xxix. doi: 10.1016/j.ajo.2018.08.038. Epub 2018 Sep 5. PMID 30194931

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the investigative sites in France, Germany, and the United States from 29 November 2017 to 29 June 2022.
Pre-assignment Details: A total of 66 unique male participants with Choroideremia were treated in the study. Of which 60 participants were treated in treatment Period 1 and 50 participants completed Period 1. 50 participants from Period 1 enrolled in Period 2 along with 6 unique participants who were treated in the first eye in a previous study (20150371 [NCT02553135], THOR-TUE-01 [NCT02671539]). 53 participants completed Period 2.
Groups:
- Treatment Period 1: BIIB111: After vitrectomy and retinal detachment in the study eye 1, participants received a single administration of BIIB111, 1 * 10^11 gp, as a sub-retinal injection on Day 0 (surgery day) of Period 1.
- Treatment Period 2: BIIB111: After vitrectomy and retinal detachment in the study eye 2, participants received a single administration of BIIB111, 1 * 10^11 gp, as a sub-retinal injection on Day 0 (surgery day) of Period 2.
Period: Treatment Period 1(Day 1 up to Month 12)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Started | 60 | 0
Completed | 50 | 0
Not Completed | 10 | 0
Not completed — Serious Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Site Terminated by Sponsor | 2 | 0
Not completed — Reason not Specified | 2 | 0
Period: Treatment Period 2 (Month13 to Month24)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Started | 0 | 56 (Note: Started population included 50 participants who completed Period 1 and 6 unique participants who were enrolled in period 2.)
Completed | 0 | 53
Not Completed | 0 | 3
Not completed — Death | 0 | 1
Not completed — Reason not Specified | 0 | 2

BASELINE CHARACTERISTICS:
Population: All Treated Subjects analysis set included all participants who completed the 'Day of Surgery' visit of Period 1 or 2. The baseline data were collected and reported for overall population of unique participants instead of period-wise treated population.
Groups:
- All Treated Participants: After vitrectomy and retinal detachment in the study eye 1 and study eye 2, participants received a single administration of BIIB111, 1 * 10^11 gp, as a sub-retinal injection on Day 0 (surgery day) of Period 1 and Period 2 respectively.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.7 (13.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 65
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Best-Corrected Visual Acuity (BCVA) as Measured by the Early Treatment of Diabetic Retinopathy Study (ETDRS) Chart in Letters at Month 12
Description: BCVA was assessed for both eyes using the ETDRS visual acuity (VA) chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. BCVA is reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters) in the study eyes. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Time Frame: Month 12
Population: All Treated Subjects analysis set included all participants who completed the 'Day of Surgery' visit of Period 1 or 2. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
letters
  Study Eye 1 | 68.0 (25.18) | 76.5 (13.78)
  Study Eye 2 | 82.3 (8.67) | 81.2 (10.82)

2. Primary Outcome: Ophthalmic Examination Assessment: Mean Intraocular Pressure (IOP) at Month 12
Description: IOP, the fluid pressure inside the eye was measured and reported in millimeters mercury (mmHg).
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 52
mmHg
  Study Eye 1 | 13.5 (3.09) | 13.5 (3.12)
  Study Eye 2 | 14.9 (2.50) | 13.5 (3.55)

3. Primary Outcome: Ophthalmic Examination Assessment: Number of Participants With Clinically Significant Abnormalities in Slit Lamp Examination
Description: Slit lamp examinations of study eyes included examination of Cornea, Conjunctiva, Iris, Lens, and Anterior Segment.
Time Frame: Baseline, Month 12
Population: All Treated Subjects analysis set included all participants who completed the 'Day of Surgery' visit of Period 1 or 2. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis of specified category at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 60 | 56
Participants
  Cornea: Study Eye 1: Baseline | 0 | 0
  Cornea: Study Eye 1: Month 12: number analyzed (Participants) | 15 | 53
  Cornea: Study Eye 1: Month 12 | 0 | 0
  Cornea: Study Eye 2: Baseline | 0 | 0
  Cornea: Study Eye 2: Month 12: number analyzed (Participants) | 15 | 53
  Cornea: Study Eye 2: Month 12 | 0 | 0
  Conjunctiva: Study Eye 1: Baseline | 0 | 1
  Conjunctiva: Study Eye 1: Month 12: number analyzed (Participants) | 15 | 53
  Conjunctiva: Study Eye 1: Month 12 | 0 | 0
  Conjunctiva: Study Eye 2: Baseline | 0 | 0
  Conjunctiva: Study Eye 2: Month 12: number analyzed (Participants) | 15 | 53
  Conjunctiva: Study Eye 2: Month 12 | 0 | 0
  Iris: Study Eye 1: Baseline | 0 | 0
  Iris: Study Eye 1: Month 12: number analyzed (Participants) | 15 | 53
  Iris: Study Eye 1: Month 12 | 0 | 0
  Iris: Study Eye 2: Baseline | 0 | 0
  Iris: Study Eye 2: Month 12: number analyzed (Participants) | 15 | 53
  Iris: Study Eye 2: Month 12 | 0 | 0
  Lens: Study Eye 1: Baseline | 2 | 2
  Lens: Study Eye 1: Month 12: number analyzed (Participants) | 15 | 53
  Lens: Study Eye 1: Month 12 | 1 | 4
  Lens: Study Eye 2: Baseline | 2 | 2
  Lens: Study Eye 2: Month 12: number analyzed (Participants) | 15 | 53
  Lens: Study Eye 2: Month 12 | 0 | 3
  Anterior Segment: Study Eye 1: Baseline | 0 | 0
  Anterior Segment: Study Eye 1: Month 12: number analyzed (Participants) | 15 | 53
  Anterior Segment: Study Eye 1: Month 12 | 0 | 0
  Anterior Segment: Study Eye 2: Baseline | 0 | 0
  Anterior Segment: Study Eye 2: Month 12: number analyzed (Participants) | 15 | 53
  Anterior Segment: Study Eye 2: Month 12 | 0 | 0

4. Primary Outcome: Ophthalmic Examination Assessment: Number of Participants With Clinically Significant Abnormalities in Dilated Ophthalmoscopy
Description: Dilated Ophthalmoscopy examination of study eyes included examination of Vitreous, Macula, Peripheral retina, Choroid, and Optic nerve.
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 60 | 56
Participants
  Vitreous: Study Eye 1: Baseline | 0 | 0
  Vitreous: Study Eye 1: Month 12: number analyzed (Participants) | 15 | 53
  Vitreous: Study Eye 1: Month 12 | 1 | 1
  Vitreous: Study Eye 2: Baseline | 0 | 0
  Vitreous: Study Eye 2: Month 12: number analyzed (Participants) | 15 | 53
  Vitreous: Study Eye 2: Month 12 | 0 | 1
  Macula: Study Eye 1: Baseline | 57 | 54
  Macula: Study Eye 1: Month 12: number analyzed (Participants) | 15 | 53
  Macula: Study Eye 1: Month 12 | 15 | 51
  Macula: Study Eye 2: Baseline | 58 | 54
  Macula: Study Eye 2: Month 12: number analyzed (Participants) | 15 | 53
  Macula: Study Eye 2: Month 12 | 15 | 51
  Peripheral Retina: Study Eye 1: Baseline | 58 | 54
  Peripheral Retina: Study Eye 1: Month 12: number analyzed (Participants) | 15 | 53
  Peripheral Retina: Study Eye 1: Month 12 | 15 | 51
  Peripheral Retina: Study Eye 2: Baseline | 58 | 54
  Peripheral Retina: Study Eye 2: Month 12: number analyzed (Participants) | 15 | 53
  Peripheral Retina: Study Eye 2: Month 12 | 15 | 51
  Choroid: Study Eye 1: Baseline | 58 | 54
  Choroid: Study Eye 1: Month 12: number analyzed (Participants) | 15 | 53
  Choroid: Study Eye 1: Month 12 | 15 | 51
  Choroid: Study Eye 2: Baseline | 58 | 54
  Choroid: Study Eye 2: Month 12: number analyzed (Participants) | 15 | 53
  Choroid: Study Eye 2: Month 12 | 15 | 51
  Optic Nerve: Study Eye 1: Baseline | 5 | 4
  Optic Nerve: Study Eye 1: Month 12: number analyzed (Participants) | 15 | 53
  Optic Nerve: Study Eye 1: Month 12 | 0 | 3
  Optic Nerve: Study Eye 2: Baseline | 6 | 4
  Optic Nerve: Study Eye 2: Month 12: number analyzed (Participants) | 15 | 53
  Optic Nerve: Study Eye 2: Month 12 | 0 | 4

5. Primary Outcome: Ophthalmic Examination Assessment: Number of Participants With Lens Opacity Grading
Description: The following lens opacity grades are reported for categories 1-4: Nuclear Opalescence grade, Nuclear Color grade, Cortical Cataract grade, and Posterior Cataract grade. Opacification severity is graded on a decimal scale, scores can range from 0.1 (no opacity) to 6.9 (maximum opacity) for the Nuclear Opalescence and Nuclear Color grades; and scores can range from 0.1 (lens clear) to 5.9 (lens unclear) for the Cortical and Posterior Cataract grades. Category 1 includes values 1, 1.0 and 0.x, Category 2 includes values 2, 2.0 and 1.x, Category 3 includes values 3, 3.0 and 2.x, and Category 4 includes values 4, 4.0, 3.x and any values above 4. For each opacification type the higher grading scores indicate greater severity.
Time Frame: Month 12
Population: All Treated Subjects analysis set included all participants who completed the 'Day of Surgery' visit of Period 1 or 2. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis of specified category of specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 50
Participants
  Nuclear Opalescence Grade: Category 1: Study Eye 1: number analyzed (Participants) | 14 | 50
  Nuclear Opalescence Grade: Category 1: Study Eye 1 | 13 | 38
  Nuclear Opalescence Grade: Category 2: Study Eye 1: number analyzed (Participants) | 14 | 50
  Nuclear Opalescence Grade: Category 2: Study Eye 1 | 1 | 8
  Nuclear Opalescence Grade: Category 3: Study Eye 1: number analyzed (Participants) | 14 | 50
  Nuclear Opalescence Grade: Category 3: Study Eye 1 | 0 | 4
  Nuclear Opalescence Grade: Category 4: Study Eye 1: number analyzed (Participants) | 14 | 50
  Nuclear Opalescence Grade: Category 4: Study Eye 1 | 0 | 0
  Nuclear Opalescence Grade: Category 1: Study Eye 2 | 14 | 38
  Nuclear Opalescence Grade: Category 2: Study Eye 2 | 1 | 10
  Nuclear Opalescence Grade: Category 3: Study Eye 2 | 0 | 2
  Nuclear Opalescence Grade: Category 4: Study Eye 2 | 0 | 0
  Nuclear Color Grade: Category 1: Study Eye 1: number analyzed (Participants) | 14 | 50
  Nuclear Color Grade: Category 1: Study Eye 1 | 14 | 41
  Nuclear Color Grade: Category 2: Study Eye 1: number analyzed (Participants) | 14 | 50
  Nuclear Color Grade: Category 2: Study Eye 1 | 0 | 5
  Nuclear Color Grade: Category 3: Study Eye 1: number analyzed (Participants) | 14 | 50
  Nuclear Color Grade: Category 3: Study Eye 1 | 0 | 4
  Nuclear Color Grade: Category 4: Study Eye 1: number analyzed (Participants) | 14 | 50
  Nuclear Color Grade: Category 4: Study Eye 1 | 0 | 0
  Nuclear Color Grade: Category 1: Study Eye 2 | 15 | 41
  Nuclear Color Grade: Category 2: Study Eye 2 | 0 | 7
  Nuclear Color Grade: Category 3: Study Eye 2 | 0 | 2
  Nuclear Color Grade: Category 4: Study Eye 2 | 0 | 0
  Cortical Cataract Grade: Category 1: Study Eye 1: number analyzed (Participants) | 14 | 50
  Cortical Cataract Grade: Category 1: Study Eye 1 | 13 | 43
  Cortical Cataract Grade: Category 2: Study Eye 1: number analyzed (Participants) | 14 | 50
  Cortical Cataract Grade: Category 2: Study Eye 1 | 1 | 5
  Cortical Cataract Grade: Category 3: Study Eye 1: number analyzed (Participants) | 14 | 50
  Cortical Cataract Grade: Category 3: Study Eye 1 | 0 | 2
  Cortical Cataract Grade: Category 4: Study Eye 1: number analyzed (Participants) | 14 | 50
  Cortical Cataract Grade: Category 4: Study Eye 1 | 0 | 0
  Cortical Cataract Grade: Category 1: Study Eye 2 | 14 | 44
  Cortical Cataract Grade: Category 2: Study Eye 2 | 1 | 6
  Cortical Cataract Grade: Category 3: Study Eye 2 | 0 | 0
  Cortical Cataract Grade: Category 4: Study Eye 2 | 0 | 0
  Posterior Cataract Grade: Category 1: Study Eye 1: number analyzed (Participants) | 14 | 50
  Posterior Cataract Grade: Category 1: Study Eye 1 | 13 | 40
  Posterior Cataract Grade: Category 2: Study Eye 1: number analyzed (Participants) | 14 | 50
  Posterior Cataract Grade: Category 2: Study Eye 1 | 0 | 6
  Posterior Cataract Grade: Category 3: Study Eye 1: number analyzed (Participants) | 14 | 50
  Posterior Cataract Grade: Category 3: Study Eye 1 | 0 | 3
  Posterior Cataract Grade: Category 4: Study Eye 1: number analyzed (Participants) | 14 | 50
  Posterior Cataract Grade: Category 4: Study Eye 1 | 1 | 1
  Posterior Cataract Grade: Category 1: Study Eye 2 | 15 | 44
  Posterior Cataract Grade: Category 2: Study Eye 2 | 0 | 6
  Posterior Cataract Grade: Category 3: Study Eye 2 | 0 | 0
  Posterior Cataract Grade: Category 4: Study Eye 2 | 0 | 0

6. Primary Outcome: Spectral Domain Optical Coherence Tomography (SD-OCT): Foveal Subfield Thickness at Month 12
Description: SD-OCT was used to assess change in foveal subfield thickness. The measurements were taken after dilation of the participant's pupil.
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microns (µ)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
microns (µ)
  Study Eye 1 | 290.7 (69.94) | 258.0 (58.20)
  Study Eye 2 | 283.8 (46.65) | 270.9 (51.66)

7. Primary Outcome: SD-OCT: Total Macular Volume at Month 12
Description: SD-OCT was used to assess change in total macular volume. The measurements were taken after dilation of the participant's pupil.
Time Frame: Month 12
Population: All Treated Subjects analysis set included all participants who completed the 'Day of Surgery' visit of Period 1 or 2. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis of specified eye.
Measure: Mean (Standard Deviation); unit: cubic millimeters (mm^3)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
cubic millimeters (mm^3)
  Study Eye 1: number analyzed (Participants) | 14 | 53
  Study Eye 1 | 6.770 (1.1384) | 6.638 (1.0934)
  Study Eye 2 | 6.903 (1.0875) | 6.741 (1.1616)

8. Primary Outcome: SD-OCT: Central Horizontal Ellipsoid Width at Month 12
Description: SD-OCT was used to assess change in central horizontal ellipsoid width. The measurements were taken after dilation of the participant's pupil.
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: microns (μ)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 14 | 47
microns (μ)
  Study Eye 1: number analyzed (Participants) | 12 | 45
  Study Eye 1 | 2346.0 (1511.67) | 1951.2 (1223.26)
  Study Eye 2 | 2230.2 (1122.89) | 1950.1 (1188.74)

9. Primary Outcome: SD-OCT: Central Ellipsoid Area at Month 12
Description: SD-OCT was used to assess change in central ellipsoid area. The measurements were taken after dilation of the participant's pupil.
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: square millimeters (mm^2)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 8 | 28
square millimeters (mm^2)
  Study Eye 1: number analyzed (Participants) | 8 | 25
  Study Eye 1 | 3.213 (2.1098) | 2.971 (1.7374)
  Study Eye 2 | 4.404 (2.2848) | 3.810 (2.5563)

10. Primary Outcome: SD-OCT: Square Root of Central Ellipsoid Area at Month 12
Description: SD-OCT was used to assess change in square root of central ellipsoid area. The measurements were taken after dilation of the participant's pupil.
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 8 | 28
mm
  Study Eye 1: number analyzed (Participants) | 7 | 25
  Study Eye 1 | 1.6980 (0.62031) | 1.6346 (0.55842)
  Study Eye 2 | 2.0331 (0.55575) | 1.8468 (0.64385)

11. Primary Outcome: SD-OCT: Choroidal Thickness at Foveal Center at Month 12
Description: SD-OCT was used to assess change in choroidal thickness. The measurements were taken after dilation of the participant's pupil.
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microns (μ)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 52
microns (μ)
  Study Eye 1 | 185.5 (81.72) | 174.2 (85.33)
  Study Eye 2 | 207.6 (85.89) | 190.2 (87.40)

12. Primary Outcome: Fundus Autofluorescence (AF): Mean Total Area of Preserved Autofluorescence at Month 12
Description: Fundus AF was used to assess the total area of preserved AF. Areas of preserved AF were identified as well-demarcated regions of relative hyper autofluorescence (hyper AF) compared with the background areas of surrounding atrophy.
Time Frame: Month 12
Population: All Treated Subjects analysis set included all participants who completed the 'Day of Surgery' visit of Period 1 or 2. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis of specified parameter.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 50
mm^2
  Study Eye 1: number analyzed (Participants) | 13 | 50
  Study Eye 1 | 7.130 (6.2326) | 8.682 (9.8972)
  Study Eye 2: number analyzed (Participants) | 15 | 49
  Study Eye 2 | 8.157 (7.4969) | 9.682 (11.0688)

13. Primary Outcome: AF: Mean Square Root of Total Area of Preserved AF at Month 12
Description: Fundus AF was used to assess the square root of total area of preserved AF. Areas of preserved AF were identified as well-demarcated regions of relative hyper AF compared with the background areas of surrounding atrophy.
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 50
mm
  Study Eye 1: number analyzed (Participants) | 13 | 50
  Study Eye 1 | 2.4358 (1.13836) | 2.6149 (1.37197)
  Study Eye 2: number analyzed (Participants) | 15 | 49
  Study Eye 2 | 2.6214 (1.17348) | 2.7550 (1.46149)

14. Primary Outcome: AF: Mean Distance From Foveal Center to Nearest Border of Preserved AF at Month 12
Description: Fundus AF was used to assess the distance from foveal center to nearest border of preserved AF.
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
mm
  Study Eye 1 | 423.133 (559.1529) | 370.245 (733.1618)
  Study Eye 2: number analyzed (Participants) | 15 | 52
  Study Eye 2 | 539.600 (602.6063) | 525.212 (688.7141)

15. Primary Outcome: Fundus Photography: Number of Participants With Retinal Pigment Epithelium (RPE) Hyperplasia as Per Severity
Description: Number of participants with RPE hyperplasia are reported for severity grades: mild, moderate, severe.
Time Frame: Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 49
Participants
  Mild: Study Eye 1 | 7 | 26
  Mild: Study Eye 2: number analyzed (Participants) | 15 | 48
  Mild: Study Eye 2 | 9 | 23
  Moderate: Study Eye 1 | 8 | 21
  Moderate: Study Eye 2: number analyzed (Participants) | 15 | 48
  Moderate: Study Eye 2 | 6 | 23
  Severe: Study Eye 1 | 0 | 2
  Severe: Study Eye 2: number analyzed (Participants) | 15 | 48
  Severe: Study Eye 2 | 0 | 2

16. Primary Outcome: Fundus Photography: Number of Participants With Retinal Arteriolar Narrowing as Per Severity
Description: Number of participants with retinal arteriolar narrowing are reported for severity grades: mild, moderate, severe.
Time Frame: Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 50
Participants
  Mild: Study Eye 1 | 13 | 37
  Mild: Study Eye 2: number analyzed (Participants) | 15 | 49
  Mild: Study Eye 2 | 12 | 36
  Moderate: Study Eye 1 | 1 | 10
  Moderate: Study Eye 2: number analyzed (Participants) | 15 | 49
  Moderate: Study Eye 2 | 2 | 10
  Severe: Study Eye 1 | 0 | 0
  Severe: Study Eye 2: number analyzed (Participants) | 15 | 49
  Severe: Study Eye 2 | 0 | 0

17. Primary Outcome: Fundus Photography: Number of Participants With Retinal Vessel Sheathing as Per Severity
Description: Number of participants with retinal vessel sheathing are reported for severity grades: mild, moderate, severe.
Time Frame: Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 49
Participants
  Mild: Study Eye 1 | 0 | 0
  Mild: Study Eye 2: number analyzed (Participants) | 15 | 48
  Mild: Study Eye 2 | 0 | 0
  Moderate: Study Eye 1 | 0 | 0
  Moderate: Study Eye 2: number analyzed (Participants) | 15 | 48
  Moderate: Study Eye 2 | 0 | 0
  Severe: Study Eye 1 | 0 | 0
  Severe: Study Eye 2: number analyzed (Participants) | 15 | 48
  Severe: Study Eye 2 | 0 | 0

18. Primary Outcome: Fundus Photography: Number of Participants With Optic Atrophy/Pallor as Per Severity
Description: Number of participants with optic atrophy/pallor are reported for severity grades: mild, moderate, severe.
Time Frame: Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 50
Participants
  Mild: Study Eye 1 | 0 | 0
  Mild: Study Eye 2: number analyzed (Participants) | 15 | 49
  Mild: Study Eye 2 | 0 | 0
  Moderate: Study Eye 1 | 0 | 0
  Moderate: Study Eye 2: number analyzed (Participants) | 15 | 49
  Moderate: Study Eye 2 | 0 | 0
  Severe: Study Eye 1 | 0 | 0
  Severe: Study Eye 2: number analyzed (Participants) | 15 | 49
  Severe: Study Eye 2 | 0 | 0

19. Primary Outcome: Fundus Photography: Number of Participants With Optic Disc Swelling as Per Severity
Description: Number of participants with optic disc swelling are reported for severity grades: mild, moderate, severe.
Time Frame: Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 50
Participants
  Mild: Study Eye 1 | 0 | 1
  Mild: Study Eye 2: number analyzed (Participants) | 15 | 49
  Mild: Study Eye 2 | 0 | 0
  Moderate: Study Eye 1 | 0 | 0
  Moderate: Study Eye 2: number analyzed (Participants) | 15 | 49
  Moderate: Study Eye 2 | 0 | 0
  Severe: Study Eye 1 | 0 | 0
  Severe: Study Eye 2: number analyzed (Participants) | 15 | 49
  Severe: Study Eye 2 | 0 | 0

20. Primary Outcome: Microperimetry: Retinal Mean Sensitivity at Month 12
Description: Microperimetry was conducted to assess retinal mean sensitivity within the macula. Retinal mean sensitivity to light was measured in decibels in multiple spots across the central and peripheral retina (entire visual field). Higher numbers (decibels) indicate higher retinal sensitivity.
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: decibels (dB)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
decibels (dB)
  Study Eye 1 | 4.05 (4.565) | 5.93 (6.991)
  Study Eye 2 | 5.41 (5.239) | 6.37 (6.720)

21. Primary Outcome: Microperimetry: Bivariate Contour Ellipse Area 63% at Month 12
Description: Microperimetry was conducted to assess bivariate contour ellipse area 63%.
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: square degrees (deg^2)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
square degrees (deg^2)
  Study Eye 1 | 7.91 (13.287) | 2.09 (4.701)
  Study Eye 2 | 1.45 (1.874) | 1.92 (5.510)

22. Primary Outcome: Microperimetry: Bivariate Contour Ellipse Area 95% at Month 12
Description: Microperimetry was conducted to assess bivariate contour ellipse area 95%.
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: deg^2
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
deg^2
  Study Eye 1 | 23.69 (39.857) | 6.27 (14.106)
  Study Eye 2 | 4.35 (5.624) | 5.76 (16.518)

23. Primary Outcome: Microperimetry: Fixation Losses (in Percentage) at Month 12
Description: Microperimetry was conducted to assess fixation losses (in percentage) which samples the optic nerve blind spot for positive responses.
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 5 | 23
percentage (%)
  Study Eye 1 | 9.0 (12.45) | 2.2 (7.20)
  Study Eye 2 | 4.0 (8.94) | 5.0 (9.17)

24. Primary Outcome: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An AE is any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug/surgical procedure, whether or not related to the investigational product or with the surgical procedure. TEAEs are defined as AEs starting on or after the day of the first surgery.
Time Frame: Day 0 (surgery) in period 1 up to last follow up visit in period 2 (approximately 2 years)
Population: All Treated Subjects analysis set included all participants who completed the 'Day of Surgery' visit of Period 1 or 2. The AEs data were collected and reported for unique participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 60 | 56
percentage of participants | 100 | 96.4

25. Primary Outcome: Number of Participants With Vector Shedding Post-treatment at Month 3
Description: Tears (for both eyes- oculus dexter [OD] and oculus sinister [OS]), blood, urine and saliva samples were collected and tested using an appropriate assay for evidence of vector shedding. Participants with positive result for vector shredding post treatment are reported.
Time Frame: Baseline, at Month 3
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 48 | 56
Participants
  Tears OD: number analyzed (Participants) | 47 | 54
  Tears OD | 0 | 0
  Tears OS: number analyzed (Participants) | 48 | 55
  Tears OS | 0 | 0
  Blood: number analyzed (Participants) | 47 | 55
  Blood | 0 | 0
  Saliva: number analyzed (Participants) | 48 | 54
  Saliva | 0 | 0
  Urine: number analyzed (Participants) | 47 | 56
  Urine | 0 | 0

26. Primary Outcome: Number of Participants With Anti-drug Antibodies Post-treatment at Month 12
Description: Participants with antibodies to the REP-1 transgenic product are reported.
Time Frame: Month 12
Population: The immunogenicity analysis set included all participants who completed the 'Day of Surgery' visit of Period 1 or 2 with baseline sample and at least one post-surgery sample evaluable for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 60 | 56
Participants | 0 | 0

27. Primary Outcome: Vital Signs: Change From Baseline in Blood Pressure at Month 12
Description: Change from baseline in Systolic and diastolic blood pressures (BP) (millimeters of mercury [mmHg]) were reported.
Time Frame: Baseline, Month 12
Population: All Treated Subjects analysis set included all participants who completed the 'Day of Surgery' visit of Period 1 or 2. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 60 | 22
mmHg
  Systolic BP: Baseline | 122.3 (14.73) | 125.4 (11.52)
  Systolic BP: Change at Month 12: number analyzed (Participants) | 14 | 22
  Systolic BP: Change at Month 12 | -7.2 (16.12) | -2.0 (10.65)
  Diastolic BP: Baseline | 78.3 (9.56) | 80.5 (6.91)
  Diastolic BP: Change at Month 12: number analyzed (Participants) | 14 | 22
  Diastolic BP: Change at Month 12 | -1.0 (11.29) | -1.9 (9.60)

28. Primary Outcome: Vital Signs: Change From Baseline in Pulse Rate at Month 12
Description: Change from baseline in pulse rate (beats per minute) were reported.
Time Frame: Baseline, Month 12
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 60 | 22
beats per minute
  Baseline | 69.8 (13.31) | 71.5 (10.91)
  Change at Month 12: number analyzed (Participants) | 14 | 22
  Change at Month 12 | 6.7 (16.41) | 0.9 (10.46)

29. Secondary Outcome: Change From Baseline in BCVA as Measured by the ETDRS Chart
Description: BCVA was assessed for both eyes using the ETDRS VA chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. BCVA is reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters) in the study eyes. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). An increase in the number of letters read correctly means that vision has improved.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
letters
  Change at Month 12: Study Eye 1 | -8.6 (24.55) | -1.3 (7.77)
  Change at Month 12: Study Eye 2 | 2.2 (2.93) | -2.2 (8.27)

30. Secondary Outcome: AF: Change From Baseline in Total Area of Preserved Autofluorescence at Month 12
Description: Fundus AF was used to assess change in total area of preserved AF. Areas of preserved AF were identified as well-demarcated regions of relative hyper autofluorescence (hyper AF) compared with the background areas of surrounding atrophy. Here negative values indicate decline in total area of preserved autofluoroscence.
Time Frame: Baseline, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 50
mm^2
  Change at Month 12: Study Eye 1: number analyzed (Participants) | 13 | 50
  Change at Month 12: Study Eye 1 | -1.158 (1.3362) | -1.502 (1.9315)
  Change at Month 12: Study Eye 2: number analyzed (Participants) | 15 | 49
  Change at Month 12: Study Eye 2 | -0.772 (0.5381) | -1.313 (1.9967)

31. Secondary Outcome: AF: Change From Baseline in Square Root of Total Area of Preserved AF at Month 12
Description: Fundus AF was used to assess change in square root of total area of preserved AF. Areas of preserved AF were identified as well-demarcated regions of relative hyper AF compared with the background areas of surrounding atrophy. Here negative values indicate decline in total area of preserved autofluoroscence.
Time Frame: Baseline, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 50
mm
  Change at Month 12: Study Eye 1: number analyzed (Participants) | 13 | 50
  Change at Month 12: Study Eye 1 | -0.1981 (0.13033) | -0.2197 (0.18111)
  Change at Month 12: Study Eye 2: number analyzed (Participants) | 15 | 49
  Change at Month 12: Study Eye 2 | -0.1345 (0.04362) | -0.1736 (0.16090)

32. Secondary Outcome: AF: Change From Baseline in Distance From Foveal Center to Nearest Border of Preserved AF at Month 12
Description: Fundus Autofluoroscence was used to assess change in distance from foveal center to nearest border of preserved autofluoroscence. Here negative values indicate decline in total area of preserved autofluoroscence.
Time Frame: Baseline, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
mm
  Change at Month 12: Study Eye 1 | -160.000 (197.9094) | -94.321 (106.4964)
  Change at Month 12: Study Eye 2 | -76.000 (71.9107) | -80.596 (135.5793)

33. Secondary Outcome: SD-OCT: Change From Baseline in Foveal Subfield Thickness at Month 12
Description: SD-OCT was used to assess change in foveal subfield thickness. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates decline in foveal subfield thickness.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microns (μ)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
microns (μ)
  Change at Month 12: Study Eye 1 | 1.7 (53.08) | -2.9 (12.02)
  Change at Month 12: Study Eye 2 | -3.5 (7.40) | -5.7 (23.96)

34. Secondary Outcome: SD-OCT: Change From Baseline in Total Macular Volume at Month 12
Description: SD-OCT was used to assess change in total macular volume. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates decline in total macular volume.
Time Frame: Baseline, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
mm^3
  Change at Month 12: Study Eye 1: number analyzed (Participants) | 14 | 53
  Change at Month 12: Study Eye 1 | -0.201 (0.2275) | -0.188 (0.1400)
  Change at Month 12: Study Eye 2 | -0.093 (0.1344) | -0.233 (0.3969)

35. Secondary Outcome: SD-OCT: Change From Baseline in the Central Horizontal Ellipsoid Width at Month 12
Description: SD-OCT was used to assess change in central horizontal ellipsoid width. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates decline in central horizontal ellipsoid width.
Time Frame: Baseline, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: microns (μ)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 14 | 44
microns (μ)
  Change at Month 12: Study Eye 1: number analyzed (Participants) | 12 | 44
  Change at Month 12: Study Eye 1 | -156.8 (185.66) | -161.5 (299.00)
  Change at Month 12: Study Eye 2: number analyzed (Participants) | 14 | 43
  Change at Month 12: Study Eye 2 | -217.5 (388.56) | -150.4 (360.87)

36. Secondary Outcome: SD-OCT: Change From Baseline in Central Ellipsoid Area at Month 12
Description: SD-OCT was used to assess change in central ellipsoid area. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates decline in central ellipsoid area.
Time Frame: Baseline, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 7 | 27
mm^2
  Change at Month 12: Study Eye 1: number analyzed (Participants) | 6 | 23
  Change at Month 12: Study Eye 1 | -0.408 (0.2184) | -0.452 (0.2776)
  Change at Month 12: Study Eye 2 | -0.466 (0.3543) | -0.369 (0.3425)

37. Secondary Outcome: SD-OCT: Change From Baseline in Square Root of Central Ellipsoid Area at Month 12
Description: SD-OCT was used to assess change in square root of central ellipsoid area. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates decline in square root of central ellipsoid area.
Time Frame: Baseline, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 7 | 27
mm
  Change at Month 12: Study Eye 1: number analyzed (Participants) | 6 | 23
  Change at Month 12: Study Eye 1 | -0.1348 (0.08110) | -0.1345 (0.06117)
  Change at Month 12: Study Eye 2 | -0.1121 (0.08193) | -0.0944 (0.09347)

38. Secondary Outcome: SD-OCT: Change From Baseline in the Choroidal Thickness at Foveal Center at Month 12
Description: SD-OCT was used to assess change in choroidal thickness. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates decline in choroidal thickness.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microns (μ)
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 52
microns (μ)
  Change at Month 12: Study Eye 1 | -12.9 (35.57) | -13.7 (30.73)
  Change at Month 12: Study Eye 2 | -9.8 (23.73) | 2.9 (23.62)

39. Secondary Outcome: Microperimetry: Change From Baseline in Retinal Mean Sensitivity at Month 12
Description: Microperimetry was conducted to assess change in retinal mean sensitivity within the macula. Retinal mean sensitivity to light was measured in decibels in multiple spots across the central and peripheral retina (entire visual field). Higher numbers (decibels) indicate higher retinal sensitivity. A negative change from baseline indicates decline in retinal sensitivity.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
dB
  Change at Month 12: Study Eye 1 | -0.79 (1.160) | -0.38 (1.931)
  Change at Month 12: Study Eye 2 | 0.15 (0.725) | -0.73 (1.435)

40. Secondary Outcome: Microperimetry: Change From Baseline in Bivariate Contour Ellipse Area 63% at Month 12
Description: Microperimetry was conducted to assess change in bivariate contour ellipse area 63%. A negative change from baseline indicates decline in bivariate contour ellipse area 63%.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: deg^2
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
deg^2
  Change at Month 12: Study Eye 1 | 4.42 (14.383) | -0.22 (6.733)
  Change at Month 12: Study Eye 2 | -0.02 (1.296) | 0.63 (5.681)

41. Secondary Outcome: Microperimetry: Change From Baseline in the Bivariate Contour Ellipse Area 95% at Month 12
Description: Microperimetry was conducted to assess change in bivariate contour ellipse area 95%. A negative change from baseline indicates decline in bivariate contour ellipse area 95%.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: deg^2
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 15 | 53
deg^2
  Change at Month 12: Study Eye 1 | 13.23 (43.125) | -0.66 (20.204)
  Change at Month 12: Study Eye 2 | -0.09 (3.866) | 1.90 (17.006)

42. Secondary Outcome: Microperimetry: Change From Baseline in Fixation Losses (in Percentage) at Month 12
Description: Microperimetry was conducted to assess change in fixation losses (in percentage) which samples the optic nerve blind spot for positive responses. A negative change from baseline indicates decline in fixation losses.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
Number analyzed (Participants) | 4 | 14
percentage
  Change at Month 12: Study Eye 1 | 5.3 (13.60) | -4.5 (11.72)
  Change at Month 12: Study Eye 2 | -6.3 (12.50) | 2.8 (7.40)

ADVERSE EVENTS:
Time Frame: Day 0 (surgery) in period 1 up to last follow up visit in period 2 (approximately 2 years)
Description: All Treated Subjects analysis set included all participants who completed the 'Day of Surgery' visit of Period 1 or 2. The AEs data were collected and reported for unique participants enrolled in the study.
Arm/Group | Treatment Period 1: BIIB111 | Treatment Period 2: BIIB111
All-Cause Mortality (participants affected / at risk) | 0/60 | 1/56
Serious Adverse Events (participants affected / at risk) | 12/60 | 8/56
Other Adverse Events (participants affected / at risk) | 59/60 | 53/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1: BIIB111 (N=60) | Treatment Period 2: BIIB111 (N=56)
Visual acuity reduced (Eye disorders) | 10 | 6
Noninfective retinitis (Eye disorders) | 2 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Choroidal neovascularisation (Eye disorders) | 1 | 0
Eye inflammation (Eye disorders) | 1 | 0
Macular hole (Eye disorders) | 0 | 1
Retinal degeneration (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Tractional retinal detachment (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1: BIIB111 (N=60) | Treatment Period 2: BIIB111 (N=56)
Conjunctival haemorrhage (Eye disorders) | 38 | 36
Anterior chamber cell (Eye disorders) | 29 | 32
Eye pain (Eye disorders) | 9 | 10
Foreign body sensation in eyes (Eye disorders) | 11 | 10
Conjunctival hyperaemia (Eye disorders) | 11 | 6
Eye irritation (Eye disorders) | 8 | 9
Vitreal cells (Eye disorders) | 7 | 4
Vitritis (Eye disorders) | 7 | 8
Ocular discomfort (Eye disorders) | 3 | 7
Visual impairment (Eye disorders) | 9 | 4
Conjunctival oedema (Eye disorders) | 6 | 3
Vision blurred (Eye disorders) | 4 | 6
Anterior chamber flare (Eye disorders) | 5 | 4
Dry eye (Eye disorders) | 2 | 6
Metamorphopsia (Eye disorders) | 2 | 5
Photopsia (Eye disorders) | 1 | 6
Visual acuity reduced (Eye disorders) | 4 | 3
Cataract (Eye disorders) | 1 | 4
Cystoid macular oedema (Eye disorders) | 1 | 4
Eye pruritus (Eye disorders) | 3 | 3
Subretinal fluid (Eye disorders) | 3 | 2
Vitreous floaters (Eye disorders) | 1 | 4
Cataract subcapsular (Eye disorders) | 1 | 3
Eyelid ptosis (Eye disorders) | 1 | 4
Ocular hypertension (Eye disorders) | 3 | 2
Nasopharyngitis (Infections and infestations) | 8 | 6
Intraocular pressure increased (Investigations) | 6 | 8
Headache (Nervous system disorders) | 7 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally, the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor's Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of the Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03507686/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT03507686/SAP_001.pdf